CLINICAL TRIAL: NCT03304275
Title: The Feasibility of Pertussis Immunization in a Canadian Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Prince Edward Island (Other)
Collaborators: The Queen Elizabeth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 6007232
Record Dates: First submitted 2017-09-25; First posted 2017-10-06 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Pertussis
Keywords: Pertussis; Vaccination; Emergency Department
MeSH Terms: conditions — Whooping Cough; Emergencies | interventions — Boostrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emergency Department vaccination group (Experimental): Pertussis (Tdap) vaccine offered/administered in the Emergency Department
  Interventions: Behavioral: Tdap
- Public Health referral group (Experimental): Public Health referral for Pertussis (Tdap) vaccine administration offered
  Interventions: Behavioral: Tdap

INTERVENTIONS:
Behavioral: Tdap — Randomized controlled trial of 2 strategies to provide adults with the Tdap vaccine
  Other Names: Boostrix

SUMMARY:
Randomized controlled trial of 2 strategies to provide adults with the Tdap vaccine to patients presenting to the emergency department. Rates of vaccination as well as effects on department efficiency will be measured.

DETAILED DESCRIPTION:
This study is a prospective randomized, controlled trial of two strategies to provide patients with the pertussis vaccine. Eligible adult patients with be offered pertussis vaccination in the Emergency Department vs. a referral to Public Health for pertussis vaccination. The effect of both strategies on triage time as well as measure of emergency department efficiency including length of stay, time to physician and left without being seen rates will be compared. At a four-month follow up, rates of pertussis vaccination will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and above
* Have not received Tdap vaccine as an adult (age 18 and above) or have not received Tdap vaccine within 10 years, or unsure of vaccination status

Exclusion Criteria:

* Acute significant illness (Canadian Triage and Acuity Scale = 1)
* Deemed "in too much distress" by triage nurse
* Acute Febrile illness
* Allergy to vaccine or vaccine components
* Pts presenting for wound care (are normally given the vaccine as part of wound care)
* Pregnancy < 26 weeks

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Rate of immunization | One day
  Rate of patients receiving Tdap vaccine

SECONDARY OUTCOMES:
Length of Stay | One day
  Length of Stay (mins, secs) for all patients presenting to the emergency. department on study days.
Left with out being seen rate | One day
  Rate of patients leaving without being seen by a physician on study days.
Time to physician | One day
  Time to be seen by emergency physician after triage (mins, secs) on study days.
Patient refusals | One day
  Reasons for patient vaccination refusal
Nursing satisfaction | One day
  Five statements rated on 5 point likert scale (strongly disagree (1) to strongly agree (5)). The immunization strategy significantly increased my workload; patient care was negatively affected by the immunization strategy; I was unable to provide the standard of care because of the immunization strategy; patient flow within the department was negatively affected by the immunization strategy; the ED should implement the immunization strategy
Additional vaccine received | One day
  Additional vaccines administered in the Public Health referral arm
Triage time | One day
  Time (in seconds) required to triage eligible patients in the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Sibley, MD, Principal Investigator — University of Prince Edward Island
Locations (1):
- Queen Elizabeth Hospital, Charlottetown, Prince Edward Island, Canada

IPD SHARING:
Plan to Share IPD: No